CLINICAL TRIAL: NCT06237179
Title: Behavioral Exercise Training to Reduce Cardiovascular Disease Risk in Men Undergoing Androgen Deprivation Therapy (EXTRA-PC)
Brief Title: Behavioral Exercise Training to Reduce Cardiovascular Disease Risk
Acronym: EXTRA-PC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23-20934; HM20028583 (Other: Virginia Commonwealth University); 1K01HL161419-01A1 (NIH)
Record Dates: First submitted 2024-01-04; First posted 2024-02-01 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer; Supportive Care
Keywords: Prostate Cancer; Supportive Care; Exercise
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training Intervention (Experimental): The exercise program (ET) is tailored to each participant depending on his initial functional capacity, cardiorespiratory fitness and strength, to achieve ≥150 moderate to vigorous physical activity
  Interventions: Behavioral: Exercise Training Intervention
- Healthy Living Education Control (Active Comparator): Educational modules delivered remotely (or manual and telephone call) in a group-based setting to approximately match contact frequency and structure with the ET arm.
  Interventions: Behavioral: Healthy Living Education

INTERVENTIONS:
Behavioral: Exercise Training Intervention — 5.1. The behavioral ET and HLE interventions will be delivered over 12 weeks. Before starting the study, men will be asked to attend one (1) in-person small group orientation to provide an overview of each intervention arm, familiarize them with web-based and smartphone applications or hard copy manuals for delivery of intervention content, exercise logs, resistance bands, and equipment for strength training.
  Other Names: Behavioral, Exercise Training
  Arms: Exercise Training Intervention
Behavioral: Healthy Living Education — During the initial 12 weeks of the study, men randomized to the HLE group will receive educational modules delivered remotely (or manual and telephone call) in a group-based setting to approximately match contact frequency and structure with the ET arm.
  Arms: Healthy Living Education Control

SUMMARY:
To test the preliminary effectiveness of a home-based exercise training (ET) intervention to improve exercise capacity (VO2 peak & 6-minute walk distance [6MWD]) among prostate cancer (PC) patients compared to controls receiving healthy living education (HLE) at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with stage II/III/IV prostate cancer
* Be currently undergoing treatment with ADT (intermittent or prolonged)
* Have completed local curative-intent treatment, including prostatectomy or definitive radiation;
* Be >40 years of age up to 85;
* Be willing to sign an informed consent with HIPAA authorization form;
* Not have any hearing or sight impairments that result in the inability to use the telephone or hear normal conversation;
* Must be able to join an intervention group by personal computer, smartphone or telephone call and should agree to recording of an interview;
* Be without any serious medical condition that precludes safe participation in an exercise program;
* Speak English

Exclusion Criteria:

* Be unable to undergo MRI (i.e., ferromagnetic materials in body, inability to lie flat, claustrophobia);
* Have contraindications to exercise testing;
* Have pre-existing overt cardiovascular disease/heart failure;
* Active illness/infection;
* Hemoglobin < 7.0 grams/dL
* Platelet count < 10 x 109/L

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-21 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in maximal exercise capacity (VO2 peak) at 12 weeks | Baseline, 12 weeks, and 24 weeks
  Exercise capacity will be measured by the maximal volume of oxygen utilization (VO2 peak) during a supine graded cardiopulmonary exercise test done in conjunction with cardiac magnetic resonance (exeCMR+CPET). VO2 will be measured in both relative (ml/kg/minute) and absolute (L/minute) terms.
Change from baseline in sub-maximal exercise capacity (6MWD) at 12 weeks | Baseline, 12 weeks, and 24 weeks
  The distance walked in a sub-maximal 6-minute walk test (6MWD). 6MWD will be reported as meters walked (m).

SECONDARY OUTCOMES:
Stroke Volume (SV) as a cardiac determinant of exercise capacity among men undergoing ADT following 12 weeks of ET vs HLE controls. | Baseline, 12 weeks
  By measuring resting and exercise -associated left ventricular (LV) end-diastolic (EDV) and end-systolic volumes (ESV) we will calculate stroke volume (SV) in milliliters/beat (ml).
  SV = EDV - ESV
Left ventricular ejection fraction (LVEF) as a cardiac determinant of exercise capacity among men undergoing ADT following 12 weeks of ET vs HLE controls. | Baseline, 12 weeks
  By measuring resting and exercise-associated stroke volumes (SV) as a proportion of end-diastolic volumes (EDV) we will calculate left ventricular ejection fraction (%).
  LVEF = SV/EDV
Cardiac output (CO) as a cardiac determinant of exercise capacity among men undergoing ADT following 12 weeks of ET vs HLE controls. | Baseline, 12 weeks
  By measuring resting and exercise-associated stroke volume (SV) and the heart rate (HR) in conjunction with image acquisition we will calculate cardiac output in liters per minute (L/min).
  CO = SV x HR
Arterial-venous oxygen (a-vO2) difference as a musculoskeletal determinant of exercise capacity among men undergoing ADT following 12 weeks of ET vs HLE controls. | Baseline, 12 weeks
  From the exercise tests we will calculate a-vO2 difference using the FICK equation. The difference in oxygen saturation between the venous circulation and the arterial circulation will be reported in milliliters (ml) and also expressed as ml/100ml of blood (%)
  a-vO2 = VO2 / CO
Change in lean body mass | Baseline, 12 weeks
  We will conduct body composition assessments using bioelectrical impedance analysis (BIA) and a Dual Energy X-Ray Absorptiometry (DXA) scan. We will use dual X-ray absorptiometry (DEXA) to assess whole body composition for lean body mass.
  Lean body mass will be reported as kilograms (kg)
Change in fat mass | Baseline, 12 weeks
  We will conduct body composition assessments using bioelectrical impedance analysis (BIA) and a Dual Energy X-Ray Absorptiometry (DXA) scan. We will use dual X-ray absorptiometry (DEXA) to assess whole body composition for fat mass as well as distribution patterns of adiposity, e.g., visceral adipose tissue.
  Fat mass and visceral fat mass will be reported in kilograms (kg) and body fat percentage will be reported as fat mass / body mass (%)
Neighborhood Environment & Walkability Survey (NEWS-A) | Baseline, 12 weeks, 24 weeks
  NEWS-A is a validated self-reported survey used to assess factors that are correlates or determinants of participants ability to engage in physical activity in their neighborhoods. For example, higher walkability is determined by availability of sidewalks and access to nearby facilities.
Change in physical activity assessed with the Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline, 12 weeks, 24 weeks
  GLTEQ is a self-report survey to determine the level typical activity a participant engages in each week. Higher scores on the index indicate more activity.
Change in physical activity assessed with Accelerometry | Baseline, 12 weeks, 24 weeks
  The ActivPAL and Actigraph accelerometers provide an objective assessment of sedentary sitting time and increasing intensities of physical activity in minutes per week
Change in self-efficacy to navigate barriers to engaging in exercise | Baseline, 12 weeks, 24 weeks
  A self report of self-efficacy to engage in exercise or physical activity under different challenging conditions such as when experiencing fatigue. Higher scores indicate increased confidence to navigate barriers.
Change in self-efficacy to walk for increasing periods of time. | Baseline, 12 weeks, 24 weeks
  A self report of self-efficacy to engage in walking for an increasing period of time. Higher scores indicate increased confidence to walk for a longer periods of time without resting.
Change in Functional Assessment of Cancer Therapy - Prostate (FACT-P) scores | Baseline, 12 weeks, 24 weeks
  FACT-P is a validated self report measures of different domains of quality of life that are important for men who have been diagnosed with prostate cancer. Subscale scores can be assessed to gauge functional wellbeing, physical wellbeing, social wellbeing and emotional wellbeing as well as prostate specific wellbeing. Higher scores indicate a higher quality of life on overall and sub scales.
Change in health-related quality of life (SF-36) scores | Baseline, 12 weeks, 24 weeks
  SF-36 (RAND) is a validated self report measure of different domains of health-related quality of life that are important for adults. Higher scores indicate a higher health-related quality of life .
Change in fatigue measured with the patient reported outcomes measurement information system (PROMIS) - Fatigue scores | Baseline, 12 weeks, 24 weeks
  PROMIS - Fatigue is a validated self-report measure of fatigue among patients diagnosed with cancer and higher scores indicate a lower level of fatigue.
Change in physical function measured with the patient reported outcomes measurement information system (PROMIS) - Physical Functioning scores | Baseline, 12 weeks, 24 weeks
  PROMIS - Physical Functioning is a validated self-report measure of physical functioning among patients diagnosed with cancer and higher scores indicate a better function.
Change in sleep disturbance measured with the patient reported outcomes measurement information system (PROMIS) - Sleep Disturbance scores | Baseline, 12 weeks, 24 weeks
  PROMIS - Sleep Disturbance is a validated self-report measure of sleep disturbance among patients diagnosed with cancer and higher scores indicate less sleep disruption.
Change in depressive symptoms measured with the patient reported outcomes measurement information system (PROMIS) - Depression scores | Baseline, 12 weeks, 24 weeks
  PROMIS - Depression is a validated self-report measure of depressive symptoms among patients diagnosed with cancer and higher scores indicate less symptoms.
Change in anxiety measured with the patient reported outcomes measurement information system (PROMIS) - Anxiety scores | Baseline, 12 weeks, 24 weeks
  PROMIS - Anxiety is a validated self-report measure of depressive symptoms among patients diagnosed with cancer and higher scores indicate less symptoms.
Change in emotional distress measured with the patient reported outcomes measurement information system (PROMIS) - Emotional Distress scores | Baseline, 12 weeks, 24 weeks
  PROMIS - Anxiety is a validated self-report measure of depressive symptoms among patients diagnosed with cancer and higher scores indicate less symptoms.
Change in fatigue measured with the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) scale | Baseline, 12 weeks, 24 weeks
  FACUT-F is a validated self-report measure of fatigue among patients undergoing treatment for a chronic illness and higher scores indicate less fatigue.
Change in perceived stress as measured with Cohen's perceived stress scale (PSS) | Baseline, 12 weeks, 24 weeks
  PSS is a validated self-report measure of perceived stress and higher scores indicate more perceived stress.
Change in physical function assessed with the Short Physical Performance Battery (SPPB) | Baseline, 12 weeks, 24 weeks
  SPPB is a validated objective assessment of 3 domains of physical function that includes gait speed, grip strength and time taken to stand from a chair 5 times. Each down is scored on a scale of 0-4 with a total score summed from each domain. A higher score is indicative of better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Lucas, PhD, Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - Richmond Veterans Affairs Medical Center, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No